CLINICAL TRIAL: NCT00101894
Title: An Open-Label, Dose-Finding Study to Evaluate the Safety of AMG 706 Plus Panitumumab Plus Chemotherapy in the Treatment of Subjects With Metastatic Colorectal Cancer
Brief Title: Safety of AMG 706 Plus Panitumumab Plus Chemotherapy in the Treatment of Subjects With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040205; NCT00107328 (obsolete NCT alias)
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Rectal Cancer; Colon Cancer
Keywords: AMG 706; Panitumumab
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Folfox protocol; motesanib diphosphate; Panitumumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (14):
- Part 2 AMG 706 (MTD) + FOLFOX-4 (Experimental): Maximum Tolerated Dose of AMG 706 established in Part 1b + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706
- 125 mg QD AMG 706 + FOLFOX-4 (Experimental): 125 mg QD AMG 706 + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706
- 50 mg QD AMG706 + panitumumab + FOLFIRI (Experimental): 50 mg QD AMG706 + panitumumab + FOLFIRI
  Interventions: Drug: AMG 706; Biological: Panitumumab (Part 1a only); Drug: FOLFIRI
- Part 2 AMG 706 (MTD) + FOLFIRI (Experimental): Maximum Tolerated Dose of AMG 706 established in Part 1b + FOLFIRI
  Interventions: Drug: AMG 706; Drug: FOLFIRI
- 100 mg QD AMG 706 + FOLFIRI (Experimental): 100 mg AMG 706 + FOLFIRI
  Interventions: Drug: AMG 706; Drug: FOLFIRI
- 75 mg QD AMG 706 + panitumumab + FOLFOX-4 (Experimental): 75 mg QD AMG 706 + panitumumab + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706; Biological: Panitumumab (Part 1a only)
- 75 mg BID AMG 706 + panitumumab + FOLFIRI (Experimental): 75 mg BID AMG 706 + panitumumab + FOLFIRI
  Interventions: Drug: AMG 706; Biological: Panitumumab (Part 1a only); Drug: FOLFIRI
- 125 mg QD AMG 706 + panitumumab + FOLFIRI (Experimental): 125 mg QD AMG 706 + panitumumab + FOLFIRI
  Interventions: Drug: AMG 706; Biological: Panitumumab (Part 1a only); Drug: FOLFIRI
- 125 mg QD AMG 706 + FOLFIRI (Experimental): 125 mg QD AMG 706 + FOLFIRI
  Interventions: Drug: AMG 706; Drug: FOLFIRI
- 100 mg QD AMG 706 + panitumumab + FOLFIRI (Experimental): 100 mg QD AMG 706 + panitumumab + FOLFIRI
  Interventions: Drug: AMG 706; Biological: Panitumumab (Part 1a only); Drug: FOLFIRI
- 75 mg QD AMG 706 + FOLFOX-4 (Experimental): 75 mg QD AMG 706 + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706
- 100 mg QD AMG 706 + FOLFOX-4 (Experimental): 100 mg QD AMG 706 + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706
- 50 mg QD AMG 706 + panitumumab + FOLFOX-4 (Experimental): 50 mg QD AMG 706 + panitumumab + FOLFOX-4
  Interventions: Drug: FOLFOX-4; Drug: AMG 706; Biological: Panitumumab (Part 1a only)
- 75 mg QD AMG706 + panitumumab + FOLFIRI (Experimental): 75 mg QD AMG706 + panitumumab + FOLFIRI
  Interventions: Drug: AMG 706; Biological: Panitumumab (Part 1a only); Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFOX-4 — The FOLFOX-4 regimen will be administered every 2 weeks as follows:
  Day 1: oxaliplatin (ELOXATIN™) 85 mg/m2 IV infusion and leucovorin racemate 200 mg/m2 (or 100 mg/m2 l-LV) IV infusion given over 120 ± 10 minutes at the same time in separate bags using a Y-line, followed by 5-FU 400 mg/m2 IV bolus given over 2 to 4 minutes, followed by 5-FU 600 mg/m2 IV infusion as a 22-hour ± 2 hours continuous infusion Day 2: leucovorin racemate 200 mg/m2 (or 100 mg/m2 l-LV) IV infusion over 120 ± 10 minutes, followed by 5-FU 400 mg/m2 IV bolus given over 2 to 4 minutes, followed
  Arms: 100 mg QD AMG 706 + FOLFOX-4; 125 mg QD AMG 706 + FOLFOX-4; 50 mg QD AMG 706 + panitumumab + FOLFOX-4; 75 mg QD AMG 706 + FOLFOX-4; 75 mg QD AMG 706 + panitumumab + FOLFOX-4; Part 2 AMG 706 (MTD) + FOLFOX-4
Drug: AMG 706 — AMG 706 is a small organic molecule that has been shown in preclinical pharmacology studies to be a potent, oral, multi-kinase inhibitor with anti-angiogenic and anti-tumor activity achieved by selectively inhibiting all known VEGF receptors, PDGF receptor, and Kit.
Biological: Panitumumab (Part 1a only) — Panitumumab will be administered by IV infusion at a dose of 6 mg/kg on day 1 of each 2-week cycle.
  Arms: 100 mg QD AMG 706 + panitumumab + FOLFIRI; 125 mg QD AMG 706 + panitumumab + FOLFIRI; 50 mg QD AMG 706 + panitumumab + FOLFOX-4; 50 mg QD AMG706 + panitumumab + FOLFIRI; 75 mg BID AMG 706 + panitumumab + FOLFIRI; 75 mg QD AMG 706 + panitumumab + FOLFOX-4; 75 mg QD AMG706 + panitumumab + FOLFIRI
Drug: FOLFIRI — Irinotecan will be administered over 90 minutes ± 15 minutes on day 1 of each 2-week cycle. Leucovorin will be administered over 2 hours ± 15 minutes during the irinotecan infusion but without mixing, immediately followed by a 5-FU bolus and a 5-FU 46-hour ± 2-hour continuous intravenous infusion.
  Arms: 100 mg QD AMG 706 + FOLFIRI; 100 mg QD AMG 706 + panitumumab + FOLFIRI; 125 mg QD AMG 706 + FOLFIRI; 125 mg QD AMG 706 + panitumumab + FOLFIRI; 50 mg QD AMG706 + panitumumab + FOLFIRI; 75 mg BID AMG 706 + panitumumab + FOLFIRI; 75 mg QD AMG706 + panitumumab + FOLFIRI; Part 2 AMG 706 (MTD) + FOLFIRI

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of AMG 706 plus panitumumab when administered with either FOLFIRI or FOLFOX4 chemotherapy regimens. This is a Phase 1b clinical study.

ELIGIBILITY:
For complete inclusion and exclusion criteria, please refer to the investigator. Inclusion Criteria

1. Competent to comprehend, sign, and date an Institutional Review Board (IRB) approved informed consent form
2. Diagnosis of metastatic colorectal adenocarcinoma (may have received 1 prior chemotherapy regimen for metastatic CRC)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate hematological function
5. Adequate renal function
6. Adequate hepatic function
7. Life expectancy of greater than or equal to 3 months as documented by the investigator

Exclusion Criteria:

1. More than 1 prior chemotherapy regimen for metastatic CRC
2. Central nervous system (CNS) metastases
3. History of venous thrombosis
4. Myocardial infarction, cerebrovascular accident, transient ischemic attack, grade 2 or greater peripheral vascular disease, congestive heart failure, ongoing arrhythmias requiring medication, or unstable angina within 1 year before study enrollment
5. History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on screening chest computed tomograph (CT) scan
6. Average systolic blood pressure > 150mm Hg or average diastolic blood pressure of > 90mm Hg
7. Radiotherapy within 28 days of study enrollment or within 14 days of study enrollment for peripheral lesions
8. Prior AMG 706, oral inhibitors of AMG706, panitumumab, or another anti-EGFr monoclonal antibody (mAb) (e.g., cetuximab [Erbitux®] or EMD 72000)
9. Systemic chemotherapy within 28 days before study enrollment
10. Major surgery within 28 days or minor surgery within 7days of study enrollment
11. History of life threatening ventricular arrhythmia (eg, sustained ventricular tachycardia)
12. Female and male subjects of childbearing potential not using adequate contraceptive precautions
13. Participation in therapeutic clinical trials within 30 days before study enrollment
14. Not recovered from all previous therapies
15. Clinically significant open would, ulcer or fracture
16. Any co-morbid medical condition that would increase the risk of toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-12; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Part 1a - The incidence of adverse events and clinical laboratory abnormalities defined as dose-limiting toxicities | First 2 cycles
Part 1b - The incidence of adverse events and clinical laboratory abnormalities defined as dose-limiting toxicities | First 2 cycles
Part 2 - The overall objective tumor response rate (complete and partial response) in subjects treated with AMG 706 (at the dose determined in Part 1b), with either the FOLFIRI or FOLFOX-4 chemotherapy regimen | Every 8 weeks (+/- 7 days)

SECONDARY OUTCOMES:
Part 1a - The PK of irinotecan (and its active metabolite SN38) when administered as a part of the FOLFIRI regimen with panitumumab and AMG 706 | Cycle 1 and 2 (Days 1, 2, 3)
Part 1a - The PK of oxaliplatin when administered as a part of the FOLFOX-4 regimen with panitumumab and AMG 706 | Cycle 1 and 2 (Day 1)
Part 1a - The objective tumor response rate (complete and partial response) throughout the study | Every 6 to 8 weeks
Part 1b - The incidence of adverse events and clinical laboratory abnormalities not defined as dose-limiting toxicities | Every visit
Part 1b - The PK of AMG 706 when administered with either the FOLFIRI or FOLFOX-4 chemotherapy regimen | Cycle 2 (Day 1-2), Cycle 3 (Day 1)
Part 1b - The PK of 5-FU when administered as a part of the FOLFIRI or FOLFOX-4 regimen with AMG 706 | Cycle 1 and 2 (Day 3)
Part 2 - Duration of response: (Calculated for only those subjects who respond) | Time from first objective tumor response (subsequently confirmed at least 4 weeks later) to objective disease progression or death.
Part 2 - Time-to-progression | Time from first dose of investigational product to objective disease progression or death due to disease progression.
Part 1b - The PK of irinotecan (and its active metabolite SN38) when administered as a part of the FOLFIRI regimen with AMG 706 | Cycle 1 and 2 (Days 1, 2, 3)
Part 1b- The PK of oxaliplatin when administered as a part of the FOLFOX-4 regimen with AMG 706 | Cycle 1 and 2 (Day 1)
Part 1b - The objective tumor response rate (complete and partial response) throughout the study | Every 8 weeks (+/- 7 days)
Part 2 - Overall survival | Time from first dose of investigational product to death. Subjects who have not died while on study or are lost to follow-up will be censored at their last contact date. (Time on study plus 36 months of long term follow-up)
Part 2 - The incidence of adverse events and clinical laboratory abnormalities | Every visit
Part 2 - The PK of AMG 706 when administered with either the FOLFIRI or FOLFOX-4 chemotherapy regimen (at a subset of the study centers with the capabilities to draw, ship and process PK samples) | Cycles 2, 4, 7, and every 3 subsequent cycles (Day 1)
Exploratory - Potential biomarker development based on assessment of blood cells, tumor cells, and urine and the proposed mechanism of action of study drugs, and response | Day 1 of cycles 1 and 2, and within 7 days of a radiographic assessment
Exploratory - The effects of genetic variation in drug metabolism genes, cancer genes, and drug target genes on subject response to investigational products (separate informed consent) | Day 1 of cycles 1 and 2, and within 7 days of a radiographic assessment
Part 2 - Progression-free survival time | Time from first dose of investigational product to objective disease progression or death, subjects who have not progressed or died while on study will be censored at their last evaluable assessment date.
Part 2 - Incidence of subjects undergoing resection of metastases for curative intent | As needed
Part 1a - The incidence of adverse events and clinical laboratory abnormalities not defined as dose-limiting toxicities | Every visit
Part 1a - The PK of AMG 706 when administered with panitumumab and either the FOLFIRI or FOLFOX-4 chemotherapy regimen | Cycle 2 (Day 1-2), Cycle 3 (Day 1)
Part 1a - The serum concentration of panitumumab when administered with AMG 706 and either the FOLFIRI or FOLFOX-4 chemotherapy regimen | Cycle 1 (Day 1), Cycle 2 (Day 1), Cycle 4 (Day 1)
Part 1a - The incidence of HAPA response following panitumumab administration | Cycle 1 (Day 1), Cycle 4 (Day 1), End of Study
Part 1a - The PK of 5-FU when administered as a part of the FOLFIRI or FOLFOX-4 regimen with panitumumab and AMG 706 | Cycle 1 and 2 (Day 3)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Tebbutt N, Kotasek D, Burris HA, Schwartzberg LS, Hurwitz H, Stephenson J, Warner DJ, Chen L, Hsu CP, Goldstein D. Motesanib with or without panitumumab plus FOLFIRI or FOLFOX for the treatment of metastatic colorectal cancer. Cancer Chemother Pharmacol. 2015 May;75(5):993-1004. doi: 10.1007/s00280-015-2694-y. Epub 2015 Mar 15. PMID 25772756
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com